CLINICAL TRIAL: NCT07369856
Title: Spot Analysis of Natriuresis to Guide up- or Down-titration of Diuretic Therapy in Ambulatory Patients With Chronic Heart Failure (SAND-HF)
Brief Title: Spot Analysis of Natriuresis to Guide up- or Down-titration of Diuretic Therapy in Ambulatory Patients With Chronic Heart Failure
Acronym: SAND-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Principal Investigator, Nathaniel Hawkins, Clinical Associate Professor, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H25-01581
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Diuretics
Keywords: heart failure; diuretics; management
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 - Natriuresis-Guided Up-Titration (Experimental): Loop diuretic doses will be up-titrated based on post-diuretic urine sodium concentration measured using a point-of-care sensor. Insufficient natriuresis (<80 mmol/L) will prompt dose escalation according to a predefined algorithm.
  Interventions: Behavioral: Natriuresis-Guided Up-Titration
- Group 1 Standard of Care (Up-Titration Control) (Other): Participants will receive usual clinical management of diuretics at the discretion of their treating physician without access to urine sodium-guided titration.
  Interventions: Other: Standard care
- Group 2 Natriuresis-Guided Down-Titration (Experimental): Loop diuretic doses will be reduced based on urine sodium levels. If urine sodium ≥80 mmol/L, the current dose will be maintained; if <80 mmol/L, dose will be reduced according to a predefined algorithm. Re-titration criteria include symptomatic weight gain >2 kg in one week.
  Interventions: Behavioral: Natriuresis-Guided Down-Titration
- Group 2 Standard Care (Down-Titration Control) (Other): Participants will receive usual care without urine sodium-guided adjustments.
  Interventions: Other: Standard care
- Group 3 Observational Cohort (Other): Participants who do not meet inclusion criteria for Groups 1 or 2 will undergo baseline urine sodium assessment and routine clinical follow-up. No study-directed titration will occur.
  Interventions: Other: Observational Follow-up

INTERVENTIONS:
Behavioral: Natriuresis-Guided Up-Titration — Diuretic dose and regimen will be increased based on post-diuretic urine sodium concentration measured by a point-of-care sensor. Insufficient natriuresis (<80 mmol/L) will prompt dose escalation using a predefined algorithm.
  Arms: Group 1 - Natriuresis-Guided Up-Titration
Other: Standard care — Participants will receive usual clinical management of loop diuretics at the discretion of the treating physician, without natriuresis-guided adjustment.
  Arms: Group 1 Standard of Care (Up-Titration Control); Group 2 Standard Care (Down-Titration Control)
Behavioral: Natriuresis-Guided Down-Titration — Loop diuretic doses will be reduced based on urine sodium levels. If urine sodium ≥80 mmol/L, the current dose will be maintained; if <80 mmol/L, dose will be reduced according to a predefined algorithm. Re-titration criteria include symptomatic weight gain >2 kg in one week.
  Arms: Group 2 Natriuresis-Guided Down-Titration
Other: Observational Follow-up — Participants who do not meet inclusion criteria for Groups 1 or 2 will undergo baseline urine sodium assessment and routine clinical follow-up. No study-directed titration will occur.
  Arms: Group 3 Observational Cohort

SUMMARY:
Heart failure is a chronic condition that causes congestion and frequent hospitalizations. Diuretic doses are usually adjusted based on clinical judgment without an objective measure of response. This study will test the feasibility of using point-of-care urine sodium measurements to guide up-titration or down-titration of loop diuretics in ambulatory patients with heart failure.

Participants will be assigned to one of three groups based on congestion status. Groups 1 and 2 will be randomized 1:1 to natriuresis-guided therapy or standard care. Group 3 will be observational. The 90-day pilot trial will evaluate feasibility, clinical outcomes, and usability of a urine sodium-guided titration strategy.

DETAILED DESCRIPTION:
Heart failure is commonly associated with sodium retention and congestion. Loop diuretics are used to relieve congestion but are typically adjusted based on symptoms and clinical judgment. Spot urine sodium concentration is an objective measure of diuretic response that may help personalize treatment. A point-of-care urine sodium sensor provides rapid results and may support effective decongestion or safe reduction of diuretics when appropriate.

This prospective, two-center pilot study includes three clinical groups:

Group 1: Up-titration cohort Patients with clinical congestion or objective evidence of congestion. These participants will be randomized 1:1 to natriuresis-guided up-titration or standard care.

Group 2: Down-titration cohort Stable, euvolemic patients who may safely reduce diuretic therapy. These participants will be randomized 1:1 to natriuresis-guided down-titration or standard care.

Group 3: Observational cohort The first 100 screened patients who do not meet criteria for Groups 1 or 2. These participants will undergo baseline assessments and routine follow-up without intervention.

Urine sodium will be measured at baseline and follow-up visits. Randomized participants will have diuretic doses adjusted based on predefined algorithms. Standard care participants will receive usual clinical management.

The primary aim is to assess feasibility, including recruitment, retention, adherence to sampling procedures, and workflow implementation. Secondary analyses will describe clinical, laboratory, and symptom-based outcomes to inform development of a larger definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of heart failure according to the Universal Definition
* Use of loop diuretics
* Residing in VCH or PHC regions

Group-specific inclusion:

Group 1: Congestion score ≥5 OR objective congestion; stable furosemide ≥1 week Group 2: NYHA I-II; congestion score <5; no recent HF hospitalization; stable furosemide ≥1 month Group 3: First 100 eligible patients not meeting criteria for Groups 1 or 2

Exclusion Criteria:

* eGFR <20 mL/min/1.73m²
* Renal replacement therapy
* High-risk clinical status requiring hospitalization
* Inability to consent or perform required urine sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Congestion Score (Group 1) | 90 Days
  Change in clinical congestion score among Group 1 participants.
Successful Down-Titration of Loop Diuretics (Group 2) | 90 Days
  Proportion of Group 2 participants who maintain a reduced loop diuretic dose without needing up-titration during follow-up.

SECONDARY OUTCOMES:
Dyspnea Visual Analogue Scale (VAS) Area Under the Curve | 90 Days
  Change in dyspnea over time measured using serial VAS assessments.
Change in KCCQ-12 Score | 90 Days
  Change in heart-failure related quality of life using the KCCQ-12.
Change in NYHA Functional Class | Baseline, 30 days, 90 days
  Change in New York Heart Association functional class.
Signs of Volume Overload | Proportion of participants with clinical signs of volume overload.
  90 Days
Change in Body Weight | 90 Days
  Change in Body weight
Loop Diuretic Use and Dose | Baseline, 30 days, 90 days
  Loop Diuretic Use and Dose at different timepoints
Guideline-Directed Medical Therapy (GDMT) Use | 90 days
  Guideline-Directed Medical Therapy (GDMT) Use
NT-proBNP Concentration | 90 days
  NT-proBNP Concentration changes
Hemoconcentration | 90 days
  Changes in hemoglobin and hematocrit.
Change in Creatinine and BUN | 90 days
  Change in Creatinine and BUN
Worsening Renal Function | 90 days
  Creatinine increase ≥100% from baseline.
Hypokalemia | 90 Days
  Frequency of potassium <3.5 mEq/L.
Urine Sodium ≥80 mmol/L (Group 1) | 90 Days
  Proportion of follow-up urine samples ≥80 mmol/L.
Point-of-Care vs Laboratory Sodium Measurement Agreement | Baseline to 90 days
  Correlation between point-of-care and laboratory urine sodium measurements.
System Usability Scale | 90 Days
  Usability of the natriuresis-guided process.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Pilot feasibility study; data not intended for reuse.